CLINICAL TRIAL: NCT00860015
Title: Alimta Plus Gemcitabine as Chemotherapy for Patients With Advanced Sarcoma: A Phase II Clinical
Brief Title: Alimta Plus Gemcitabine for Advanced Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB4160
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alimta/Gemcitabine (Experimental): IV administration of drugs for 14 days for up to 4 cycles
  Interventions: Drug: Alimta; Drug: Gemcitabine

INTERVENTIONS:
Drug: Alimta — 500 mg/m2 via IV over 10 minutes
  A chemotherapy drug with indications to treat pleural mesothelioma and non-small cell lung cancer.
  Other Names: Pemetrexed
Drug: Gemcitabine — 1000 mg/m2 via IV over 90 minutes
  A nucleoside analog used as chemotherapy.
  Other Names: Gemzar

SUMMARY:
In patients with unresectable soft tissue sarcoma, what is the response rate if treated with Alimta and gemcitabine?

DETAILED DESCRIPTION:
Soft tissue sarcomas represent 0.7% of all malignancies diagnosed in the United States. The peak incidence occurs in children and young adults with a second peak occurring in middle age, resulting in significant morbidity and mortality in young, productive individuals. Although limb preserving surgery and radiation therapy have improved the primary treatment of these tumors, the therapy of advanced, metastatic tumors is unsatisfactory. The purpose of this phase II study is to evaluate the efficacy of treatment with Alimta and gemcitabine given on day 1 of a 14 day cycle to patients with unresectable or metastatic soft tissue sarcomas. Gemcitabine is an established salvage therapy for soft tissue sarcomas in combination with docetaxel. Alimta is a multitargeted antifolate drug which inhibits several folate dependent enzymes required for cell proliferation. Alimta has shown efficacy in several solid tumor types both as a single agent and in combination with other agents. The combination of Alimta and gemcitabine is synergistic and is likely to have efficacy against soft tissue sarcomas. The primary objective of this study is to determine the response rate among patients with unresectable soft tissue sarcoma treated with this combination. Secondary endpoints will evaluate the median survival of this patient population, as well as time to objective tumor response, time to treatment failure and overall survival. The toxicities of this regimen in this population will also be analyzed. Given the desperate need for new agents to treat these patients, a phase II trial of this combination therapy should be pursued.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven soft tissue sarcoma (except the following histologies: gastrointestinal stromal tumors (GIST), Kaposi's Sarcoma, mesotheliomas).
* Age ≥ 18 years
* Recurrent or progressive disease defined as an increase in size of any existing tumor mass, or the development of new tumor mass or masses, which is not amenable to definitive surgical therapy.
* Patients may have had another cancer but there must be convincing clinical evidence that the sarcoma is the disease requiring therapeutic intervention. (i.e. Several sarcoma patients have had had a prior cancer [Hodgkin's disease or breast cancer] treated years previously and then developed a clinically active sarcoma.)
* Patients may have received no prior chemotherapy, or may have failed 0-2 prior cytotoxic regimens.
* Measurable disease defined as lesions that can be measured in at least one dimension by physical examination or by means of medical imaging techniques. Ascites and pleural effusions will not be considered measurable disease.
* Karnofsky performance status of greater than or equal to 60%.
* At least 3 weeks since prior chemotherapy or at least 6 weeks since prior radiation therapy.

Exclusion Criteria:

* Soft tissue sarcomas with the following histologies: gastrointestinal stromal tumors (GIST), Kaposi's sarcoma, mesotheliomas.
* Active or uncontrolled infection
* Prior treatment with gemcitabine or Alimta
* Pregnant or lactating women
* Uncontrolled central nervous system metastases
* Inability to stop treatment with NSAIDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-08; Primary Completion 2009-08 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Taub, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Alimta/Gemcitabine: IV administration of drugs for 14 days for up to 4 cycles
  Alimta: 500 mg/m2 via IV over 10 minutes
  A chemotherapy drug with indications to treat pleural mesothelioma and non-small cell lung cancer.
  Gemcitabine: 1000 mg/m2 via IV over 90 minutes
  A nucleoside analog used as chemotherapy.
Period: Overall Study
Arm/Group | Alimta/Gemcitabine
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alimta/Gemcitabine
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  18-65 years | 10
  > 65 years | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females | 8
  Males | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1
  Hispanic | 8
  Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Tumor Best Response Rate
Description: The best response rate will include patients with both Complete Response and Partial Response after 2 months of treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Two months
Measure: Count of Participants; unit: Participants
Arm/Group | Alimta/Gemcitabine
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: Two months
Arm/Group | Alimta/Gemcitabine
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alimta/Gemcitabine (N=12)
Infection (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was deemed as closed/completed early as none of the initial 12 patients treated responded to treatment with alimta/gemcitabine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes